CLINICAL TRIAL: NCT02471469
Title: Personalizing Enzalutamide Therapy by Understanding the Relation Between the Decrease in the Expression Profile of a Panel of Preselected microRNAs, Tumor Related mRNAs and Treatment Response in Chemotherapy Naive Patients With mCRPC
Brief Title: Personalizing Enzalutamide Therapy by Understanding the Relation Between Tumor mRNAs, miRNAs and Treatment Response
Acronym: ILUMINATE
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: AKF UMCN 14.17
Record Dates: First submitted 2015-04-14; First posted 2015-06-15 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Enzalutamide, 160mg, 40 mg soft capsules, once daily — Exclusively determine pharmacokinetics and pharmacodynamics of enzalutamide for the indication according to the drug label

SUMMARY:
The primary aim is to show whether a reduction in tumor related mRNAs and a panel of selected miRNAS can be used to personalize enzalutamide therapy.

Furthermore the aim is to explore the relation between drug exposure and the decrease in the selected biomarkers and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with chemotherapy naive metastatic castration resistant prostate cancer*
* Age at least 18 years
* Patients from who it is possible to collect blood samples
* Patient who are able and willing to give written informed consent prior to screening and enrollment
* Life expectancy of > 6 months
* Measurable disease *definition of CRPC according to EAU guidelines 2014

Exclusion Criteria:

* None The study objective is to explore the effect of enzalutamide on biomarker exposure in a group of patients treated with enzalutamide in agreement with the drug label. Therefore no strict exclusion criteria will be used in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chemotherapy naive patients with metastatic CRPC
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Relation between biomarker response and therapeutic response | 6 months

SECONDARY OUTCOMES:
Relation between drug exposure, biomarker and therapeutic response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nielka van Erp, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Radboud UMC, Nijmegen
  - Canisius Wilhelmina Ziekenhuis, Nijmegen

REFERENCES:
- [Result] Benoist GE, van Oort IM, Boerrigter E, Verhaegh GW, van Hooij O, Groen L, Smit F, de Mol P, Hamberg P, Dezentje VO, Mehra N, Gerritsen W, Somford DM, van Erp NPH, Schalken JA. Prognostic Value of Novel Liquid Biomarkers in Patients with Metastatic Castration-Resistant Prostate Cancer Treated with Enzalutamide: A Prospective Observational Study. Clin Chem. 2020 Jun 1;66(6):842-851. doi: 10.1093/clinchem/hvaa095. PMID 32408351
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/32408351/